CLINICAL TRIAL: NCT01442558
Title: Comparison of Quality of Supraclavicular, Infraclavicular and Axillary Approach of Ultrasound-guided Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0081-2011-HYMC
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: relief; Intra-operative
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SCL (Active Comparator): Supraclavicular ultrasound-guided brachial plexus block
  Interventions: Drug: Bupivacaine
- ICL (Active Comparator): Infraclavicular ultrasound-guided brachial plexus block
  Interventions: Drug: Bupivacaine
- AX (Active Comparator): Axillary ultrasound-guided brachial plexus block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 5 mg/cc with adrenaline 5 mcg/cc will be injected with complete spread of the drug around nerves.

SUMMARY:
The aim of this study is to compare the quality of 3 methods of ultrasound-guided brachial plexus blocks for surgical anesthesia

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III physical status
* Surgery of distal arm, forearm or hand

Exclusion Criteria:

* Skin infection near block injection site
* Allergy to local anesthetics
* Peripheral neuropathy upper limb
* INR of more than 1.4
* Thrombocytopenia
* Opioid dependency
* Chronic pain syndrome
* Lack of orientation to person, place and time
* Patient refusal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Quality of 3 different approaches to brachial plexus block | Immediate
  Whether or not there is need for additional analgesic drugs or need to switch to general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Stav A, Reytman L, Stav MY, Portnoy I, Kantarovsky A, Galili O, Luboshitz S, Sevi R, Sternberg A. Comparison of the Supraclavicular, Infraclavicular and Axillary Approaches for Ultrasound-Guided Brachial Plexus Block for Surgical Anesthesia. Rambam Maimonides Med J. 2016 Apr 19;7(2):e0013. doi: 10.5041/RMMJ.10240. PMID 27101216